CLINICAL TRIAL: NCT02694315
Title: Comparison Between Sonographic Cervical Length and Bishop Score in Preinduction Cervical Assessment Prior to Induction of Labor as Regards Induction Success
Brief Title: Cervical Length and Bishop Score in Preinduction Cervical Assessment Prior to Induction of Labor
Status: Completed | Type: Observational
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Amr Ahmed Mahmoud Riad, Lecturer of obstetrics and gynecology, Ain Shams Maternity Hospital
Other Study IDs: sonographic cervical length
Record Dates: First submitted 2016-02-23; First posted 2016-02-29 (Estimated); Results first posted 2016-11-07 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-09

CONDITIONS: Cervical Dystocia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Induction of labor: 200 women all are primigravida between 37-42 weeks gestation to whom induction of labor will be carried out in the casualty of Ain Shams University Maternity Hospital. All participants will have an assessment of the cervix by both Bishop score system and transvaginal measurement of cervical length.
  Interventions: Other: Bishop score; Other: cervical length

INTERVENTIONS:
Other: Bishop score — calculation of modified Bishop score in numbers by digital vaginal examination
Other: cervical length — measuring cervical length by trans-vaginal ultrasound

SUMMARY:
Comparison between Sonographic Cervical Length and Bishop Score in Preinduction Cervical Assessment prior to induction of labor as regards induction success.

DETAILED DESCRIPTION:
Type of the study:

assessment of accuracy of diagnostic test.

Study setting:

The study will be performed at Ain Shams university Maternity hospital on nulliparous women at term admitted to causality for induction of labor.

Study population:

The study will be held on 200 women all are primigravida between 37-42 weeks gestation to whom induction of labor will be carried out in the casualty of Ain Shams University Maternity Hospital.

All patients will have cervical assessment by modified Bishop score and cervical length measurement by ultrasound.

Plan for induction of labor:

* Detailed and careful history will be taken from the participants as follows:

  1. Personal history: including name, age, occupation, residence and special habits of medical importance.
  2. Obstetric history: including gestational age and regular antenatal care.
  3. Past history: including any medical disorder e.g Diabetes mellitus, hypertension or any surgical procedure.
  4. History of present pregnancy: duration of pregnancy from last menstrual period, any complications occurred or any medication used during pregnancy.
* Examination of the participants:

  1. General examination: level of consciousness, vital data, complexion.
  2. Abdominal examination: fundal level, lie of the fetus, detection of any uterine contractions and fetal heart rate.
  3. Pelvic Examination : presenting part, presence of ruptured membranes and cervical assessment as regard cervical dilation, effacement, station and presenting part to calculate the modified Bishop Score.
* Investigations: complete blood count, blood group, non stress test.
* All women will have trans-vaginal ultrasound sound for assessment of cervical length.
* Protocol of trans-vaginal ultrasound will be as follows:

  1. Patient will be asked to void.
  2. Vaginal probe will be inserted using direct visualization.
  3. Identification of bladder and fetal presenting part.
  4. Identification of abnormal findings as placenta previa or absence of fetal heart motion.
  5. Identification of mid-line sagittal plane of the cervix and looking in the proximal one third of the image for the internal cervical os then pulling back the probe until the lightest touch provides good image of the cervical canal and moving the probe slightly to get the best long axis of the cervix then measuring the cervical length three times by placing the calibers appropriately and recording the distance between internal and external os then at last recording the measurement of the best image .
* If cervical length assessed by trans-vaginal ultrasound is less than 28 mm or modified Bishop Value is less than 7, the patient will receive 3mg prostaglandin E2 for pre-induction cervical ripening to be repeated after 6 hours with maximum of 2 doses. If failed cervical ripening, Cesarean section will be done.
* All Patients will be tested by antepartum fetal heart monitoring "Non stress test".This will be considered reactive if there are two or more fetal heart rate accelerations peaking at least by 15 beats/min above the baseline and lasting for 15 seconds or more from baseline, within a 20 minutes period, with or without fetal movement felt by the mother. A non-reactive tracing will be one without sufficient fetal heart rate accelerations over a 40 minutes period. Any patient with non-reassuring non stress test will be excluded.
* Successful induction will be defined as vaginal delivery within 24 hours.
* Failed induction after 24 hours will indicate lower segment cesarean section. Failed induction will be defined as an inability to achieve the active phase of labor corresponding to a cervical dilatation ≥4 cm within 12 hours of initiating oxytocin. Failure of progress was defined as no cervical dilatation during the active phase of labor for at least 2 hours or no descent of the fetal head during the second stage of labor for at least 1 hour despite adequate uterine contraction. This will be considered an indication for cesarean delivery.
* No further induction agent will be given when uterine contractions reach frequency of three in ten minutes each lasting 30-60 seconds with cervical changes. Amniotomy and oxytocin augmentation will begin when cervical dilation becomes > 3 cm.
* Oxytocin infusion will be prepared by placing 5 IU ampoule in 500 ml Ringer or Saline to achieve concentration of 10 ml\minute.
* The rate of infusion will be started at a rate of 5 miu/ml (about 10 drops per minute) and will be increased at same increment every 20 minutes according to uterine contractions.
* When the patient become in the active phase of labor, vaginal examination will be repeated every 1-2 hours to know the rate of cervical dilation.
* If patient requests pain relieve, epidural analgesia will be used.
* Fetal heart rate will be recorded every half an hour.
* Labor progress will be plotted on partogram.

ELIGIBILITY:
Inclusion Criteria:

1. Nulliparous patients.
2. Singleton pregnancy.
3. Living fetus with cephalic presentation.
4. Absence of labor pain.
5. Gestational age 37-42 weeks.
6. No previous uterine surgical procedures.
7. No Liquor abnormalities.
8. Fetal weight less than 4 kilograms.

Exclusion Criteria:

1. Non-vertex presentation.
2. Previous uterine surgery.
3. Multiple pregnancy.
4. Fetal or maternal complications that might cause cesarean section.
5. Liquor abnormalities.
6. Fetal weight more than 4 kilograms.
7. Abnormal umbilical artery Doppler indices or non-stress test.
8. Asthmatic patients or women with allergy to prostaglandins.

Ages: 17 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 200 women all are primigravida between 37-42 weeks gestation to whom induction of labor will be carried out in the casualty of Ain Shams University Maternity Hospital
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams maternity hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Induction of Labor
Started | 200
Completed | 200
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Raslan et al., 2013 reported accuracy of cervical length or Bishop score was 72% vs 63%. So, proportion of discordant pairs is 0.37. A sample of 200 would achieve a power of 80% to detect statistical significance for an effect size equivalent to odds ratio of 1.9. Two sided McNemar test was used with a confidence level 95%.
Arm/Group | Induction of Labor
Number analyzed (Participants) | 200
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 23.5 [21 to 27]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 200
  Male | 0
Gestational age [Median (Inter-Quartile Range); unit: weeks] | 39.8 [38.2 to 40.4]
Previous abortions [Number; unit: participants]
  no abortions | 173
  one abortion | 22
  two abortions | 4
  three abortions | 1
Indication of induction of labor [Number; unit: participants]
  severe pre-eclampsia | 8
  mild pre-eclampsia | 11
  intrauterine growth restriction | 3
  oligohydramnios | 17
  postdate | 89
  term rupture of membranes | 72
Need for oxytocin [Number; unit: participants]
  needed oxytocin | 116
  did not need oxytocin | 84
Outcome of induction of labor [Number; unit: participants]
  successful vaginal delivery | 114
  need for cesarean section | 86

OUTCOME MEASURES:

1. Primary Outcome: Cervical Length Prior to Labor Induction
Description: median cervical length measured by transvaginal ultrasound in centimetres
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: centimetres
Arm/Group | Induction of Labor
Number analyzed (Participants) | 200
centimetres
  successful induction of labor | 2.9 [2.8 to 3.1]
  failed induction of labor | 3 [2.8 to 3.2]

2. Primary Outcome: Bishop Score Prior to Induction of Labor
Description: median Bishop score assessed by digital vaginal examination as follows:
  1. Cervical dilatation in centimeters will be given a score of zero if closed, a score of 1 if 1-2 cm dilated, a score of 2 if 3-4 cm dilated and a score of 3 if 5 cm or more dilataion.
  2. Effacement of the cervix will be given a score of zero if 0-30%, a score of 1 if 40-50%, a score of 2 if 60-70% and a score of 3 if 80% or more.
  3. Station of fetal head will be given a score of zero if -3, a score of 1 if -2, a score of 2 if -1 to zero and a score of 3 if 1 or more.
  4. Consistency of the cervix will be given a score of zero if firm, a score of 1 if medium and a score of 2 if soft.
  5. Position of the cervix will be given a score of zero if posterior, a score of 1 if mid position and a score of 2 if anterior. So, a total score (sum of all scores) of zero at a minimum to 10 at a maximum can be estimated.
  Note that a score more than 10 means patient is in labor not needing induction of labor.
Time Frame: 72 hours
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Induction of Labor
Number analyzed (Participants) | 200
units on a scale
  successful induction of labor | 4 [3 to 5]
  failed induction of labor | 3 [3 to 4]

ADVERSE EVENTS:
Time Frame: All participants and their livebirths were followed for 72 hours following delivery for adverse events
Arm/Group | Induction of Labor
Serious Adverse Events (participants affected / at risk) | 0/200
Other Adverse Events (participants affected / at risk) | 19/200
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction of Labor (N=200)
low APGAR score (Pregnancy, puerperium and perinatal conditions) | 10 (10) — neonatal APGAR score less than 7
low birth weight (Pregnancy, puerperium and perinatal conditions) | 1 (1) — fetal birth weight less than 2500 grams
neonatal ICU admission (Pregnancy, puerperium and perinatal conditions) | 5 (5) — number of neonates admitted in neonatal ICU
maternal traumatic birth injury (Pregnancy, puerperium and perinatal conditions) | 3 (3) — any trauma in the birth tract related to delivery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No